CLINICAL TRIAL: NCT07000383
Title: Evaluation of the Efficacy and Safety of Gelsectan in the Treatment of Diarrhea-predominant Irritable Bowel Syndrome at University Medical Center Ho Chi Minh City, Vietnam: a Randomized, Open-label Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Gelsectan in the Treatment of Diarrhea-predominant Irritable Bowel Syndrome
Acronym: GELIBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHYD612025
Record Dates: First submitted 2025-05-30; First posted 2025-06-02 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome; Irritable Bowel Syndrome of Diarrhea Type (IBS-D)
Keywords: Irritable Bowel Syndrome; Gelsectan; Diarrhea-Predominant Irritable Bowel Syndrome; IBS-D; Irritable Bowel Syndrome of Diarrhea type; Xyloglucan; GELIBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Parasympatholytics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of three parallel groups: (1) Gelsectan monotherapy, (2) Gelsectan combined with an antispasmodic agent, and (3) antispasmodic therapy alone. Each participant will remain in their assigned group for the full two-month duration of the study, with assessments conducted at baseline, one month, and two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gelsectan Monotherapy (Experimental): Participants receive Gelsectan alone, administered as 2 capsules in the morning and 2 capsules in the evening during the first month; then 1 capsule in the morning and 1 in the evening during the second month.
  Interventions: Device: Gelsectan
- Gelsectan + Antispasmodic (Experimental): Participants receive Gelsectan as above, combined with a standard dose of an antispasmodic agent for 8 weeks.
  Interventions: Device: Gelsectan; Drug: Antispasmodic Agent
- Antispasmodic Only (Active Comparator): Participants receive only an antispasmodic agent (without Gelsectan) for a total duration of 8 weeks.
  Interventions: Drug: Antispasmodic Agent

INTERVENTIONS:
Device: Gelsectan — Gelsectan is a medical device containing xyloglucan, pea protein, and tannins, administered orally. Dosage: 2 capsules BID during Month 1, followed by 1 capsule BID during Month 2.
  Other Names: Xyloglucan; XG-PPT-XOS
  Arms: Gelsectan + Antispasmodic; Gelsectan Monotherapy
Drug: Antispasmodic Agent — An oral antispasmodic medication, prescribed according to standard clinical practice for IBS-D.
  Other Names: Antispasmodic drug
  Arms: Antispasmodic Only; Gelsectan + Antispasmodic

SUMMARY:
This clinical study aims to investigate the effectiveness and safety of Gelsectan, a treatment containing xyloglucan, in adults diagnosed with diarrhea-predominant irritable bowel syndrome (IBS-D) in Vietnam. IBS-D is a common digestive disorder that causes frequent diarrhea along with abdominal pain and bloating, significantly affecting patients' daily life and wellbeing.

The main goal of the study is to determine whether Gelsectan can reduce the severity of symptoms such as diarrhea, abdominal discomfort, and bloating, and improve patients' quality of life. Participants will be randomly assigned to receive either Gelsectan alone, Gelsectan combined with an antispasmodic medication, or antispasmodic medication alone. The treatment will last for two months, with regular monitoring of symptom changes and any side effects.

The investigators hypothesize that Gelsectan treatment will lead to better symptom relief and quality of life compared to standard antispasmodic treatment. The study will also carefully observe the safety profile of Gelsectan during the treatment period.

Results from this study will provide important information about the potential benefits and risks of Gelsectan for Vietnamese patients with IBS-D and may contribute to improving treatment options for this condition in Vietnam.

DETAILED DESCRIPTION:
Diarrhea-predominant irritable bowel syndrome (IBS-D) is one of the most common subtypes of IBS, accounting for approximately 30-40% of all IBS cases. In developed countries, xyloglucan-the main component of Gelsectan-has been demonstrated in various studies to be a promising therapeutic option for IBS-D. Xyloglucan forms a biofilm that protects the intestinal mucosa, reduces permeability, and helps prevent the effects of inflammatory agents and functional disturbances in the gut. Clinical studies have shown that xyloglucan not only alleviates symptoms such as diarrhea, abdominal pain, and bloating, but also restores intestinal function and significantly improves the quality of life in patients with IBS-D. IBS-D is also prevalent in Vietnam; however, there is currently no published research evaluating the use of Gelsectan for the treatment of this condition in the Vietnamese population.

This study aims to evaluate the efficacy of Gelsectan in the treatment of diarrhea-predominant irritable bowel syndrome (IBS-D) by assessing improvements in diarrhea, bloating, abdominal pain, and quality of life after 1 and 2 months of treatment. Additionally, the study investigates the safety profile of the product based on the frequency and severity of adverse events recorded throughout the intervention period.

This study is an open-label, randomized controlled clinical trial conducted at the Gastroenterology Outpatient Clinic of the University Medical Center Ho Chi Minh City, from April 2025 to April 2026. The study population includes patients aged 18 years and older, diagnosed with diarrhea-predominant irritable bowel syndrome (IBS-D) according to the Rome IV criteria.

After providing informed consent, participants will be randomly assigned to one of three intervention groups: (1) Gelsectan monotherapy, (2) Gelsectan combined with an antispasmodic agent, and (3) antispasmodic therapy alone. The intervention period lasts two months, with clinical assessments conducted at baseline, after one month, and after two months of treatment. The variables recorded include clinical remission status, number of daily diarrhea episodes, intensity of abdominal pain and bloating, and quality of life scores. Adverse events will be continuously monitored and recorded according to their severity and their relationship to the intervention.

The results of this study will provide additional clinical evidence on the efficacy and safety of Gelsectan in the treatment of IBS-D, contributing to the expansion of therapeutic options in Vietnam. The application of Gelsectan may offer practical benefits in alleviating symptoms, improving patients' quality of life, and reducing healthcare costs associated with the management and treatment of IBS-D.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of IBS-D based on the Rome IV criteria,8 including:

  * Recurrent abdominal pain occurring at least one day per week in the last three months, associated with at least two of the following: related to defecation, associated with a change in stool frequency, or associated with a change in stool form. These criteria must have been present during the last three months, with symptom onset at least six months prior to diagnosis;
  * More than 25% of bowel movements with stool types 6 or 7 and less than 25% with stool types 1 or 2 according to the Bristol Stool Form Scale.
* Signed informed consent for study participation

Exclusion Criteria:

* Pregnant or breastfeeding women
* Known allergy to any component of the study medication
* Diagnosed with diabetes mellitus
* Patients with severe comorbidities or psychiatric disorders that impair their ability to complete questionnaires or attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission of IBS-D symptoms | 1 month and 2 months
  Defined as the resolution of diarrhea, measured as ≤ 2 bowel movements per day with stool consistency < 5 on the Bristol Stool Form Scale, assessed at 1 and 2 months after treatment initiation.

SECONDARY OUTCOMES:
Incidence of adverse events | Continuous monitoring over 2 months
  Number and severity of treatment-related and unrelated adverse events reported throughout the 2-month intervention period.
IBS Severity Scoring System (IBS-SSS) | 1 month and 2 months
  The Irritable Bowel Syndrome Severity Scoring System (IBS-SSS) is used to evaluate changes in symptom severity from baseline to Month 1 and Month 2. The IBS-SSS includes five items assessing abdominal pain severity and frequency, bloating, dissatisfaction with bowel habits, and interference with life.
  Minimum score: 0; Maximum score: 500; Interpretation: Higher scores indicate worse symptom severity. Severity categories are defined as: Mild: 75-<175; Moderate: 175-<300; Severe: ≥300. A reduction of ≥50 points from baseline is considered a clinically significant improvement.
IBS-related quality of life (IBS-QoL) score | 1 month and 2 months
  The "Irritable Bowel Syndrome - Quality of Life (IBS-QoL) Questionnaire" includes 34 items across 8 domains and generates a total score ranging from 0 to 100. Interpretation: Higher scores indicate better quality of life.Total scores are categorized as follows: Very poor (<50), Poor (50-<70), Fair (70-<90), Good (90-100)

OTHER OUTCOMES:
Bloating severity | 1 month and 2 months
  Measured on a 7-point Likert scale at baseline, 1 month, and 2 months.
Abdominal pain intensity | 1 month and 2 months
  Measured on a 7-point Likert scale at baseline, 1 month, and 2 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ho Chi Minh City, Ho Chi Minh City, District 5, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided